CLINICAL TRIAL: NCT02613078
Title: Gut-Directed Hypnotherapy vs. Probiotics in Children and Adolescents With Irritable Bowel Syndrome and Functional Abdominal Pain - A Pilot Study
Brief Title: Hypnotherapy vs. Probiotics in Children With IBS and Functional Abdominal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: SymbioPharm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDG 082015
Record Dates: First submitted 2015-10-23; First posted 2015-11-24 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Irritable Bowel Syndrome; Functional Abdominal Pain Syndrome
Keywords: Children; Functional Abdominal Pain Syndrome; Irritable Bowel Syndrome; Gut-Directed Hypnotherapy; Probiotic
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Dietary Supplements; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gut-Directed Hypnotherapy (GDH) (Experimental): Gut-Directed Hypnotherapy on a daily basis (20 min each day, at least 4 times/week)
  Interventions: Behavioral: Gut-Directed Hypnotherapy; Behavioral: Self-Monitoring
- Probiotic (NS) (Experimental): Nutritional supplement SymbioLact B once a day diluted in water or tea
  Interventions: Dietary Supplement: Nutritional Supplement; Behavioral: Self-Monitoring
- Active Controls (AC) (Active Comparator): AC group keeps a symptom dairy (self-monitoring)
  Interventions: Behavioral: Self-Monitoring

INTERVENTIONS:
Behavioral: Gut-Directed Hypnotherapy — Hypnotherapy protocol is based on the Manchester protocol for gut-directed hypnotherapy and was adapted for children and adolescents. It consists of elements aiming at relaxation and suggestions for control and relief from pain and discomfort. The hypnotherapy will be provided using a CD. Children of the hypnotherapy condition will be instructed to practice with their CD on a daily basis (20 min each day, at least 4 times/week) during 4 weeks
  Arms: Gut-Directed Hypnotherapy (GDH)
Dietary Supplement: Nutritional Supplement — SymbioLact® B a preparation of Bifidobacterium lactis and vitamin B7, Biotin. Number of living organisms in one dose is at least 1 x 10^9 cfu. SymbioLact® B will be used in the dose recommended in the pediatric patient information sheet - one dose of SymbioLact® B diluted in water or tee once a day together with a main meal during 4 weeks
  Other Names: SymbioLact B
  Arms: Probiotic (NS)
Behavioral: Self-Monitoring — Use of symptom diary that questions about main bowel complains (including pain or discomfort) during the day. Applied on a daily basis (about 2 min in the evening)

SUMMARY:
Current study aims to investigate the influence of gut-directed hypnotherapy and probiotic nutritional supplement (SymbioLact B) on gastrointestinal symptoms in children with functional abdominal pain or irritable bowel syndrome compared to self-observation only. The study also includes collection of psychometric data (emotional and behavioral problems, pain coping strategies), data on activity of the autonomous nerve system as measured by heart rate variability and data on stress response (saliva cortisol levels).

DETAILED DESCRIPTION:
Children with irritable bowel syndrome (IBS) or other pain-related functional gastrointestinal disorders (FGIDs) such as functional abdominal pain (FAP) represent a considerable part of visits to pediatric practitioners. These disorders do not only decrease the quality of life but also increase the risk of symptom persistence and comorbid mental issues in adulthood. As etiology and pathophysiology of FGIDs are still a matter of research, several approaches of managing of FGIDs are commonly used: dietary interventions, probiotics, drug treatment, psychosocial interventions. While recent meta-analyses showed almost no favorable effects of dietary interventions and drug treatments (5-HT4 receptor agonists, antispasmodic and anti-diarrheal agents, antibiotics) in children with FGIDs, probiotics and psychosocial interventions remain promising regarding effective symptom relief. Several randomized controlled trials (RCT) have shown a beneficial effect of both gut directed hypnosis (GDH) and probiotics. To our knowledge, there are no studies that investigated both types of intervention in comparison to a control group intervention. This study aims to fill this gap.

In a prospective randomized study the investigators aim to obtain preliminary results about the impact of gut-directed hypnotherapy (GDH) modified for self-practicing and probiotic nutritional supplement (NS) on symptoms in children with pain-related FGIDs (IBS and FAP). This is going to be measured by the mean of number of days the children experience no abdominal pain or discomfort. Beside that the investigators plan to obtain data on abdominal pain intensity and duration and about the effects of above mentioned interventions on children's health-related quality of life (KINDL-R), pain-related disability (P-PDI), their coping abilities (PPCI) and behavioural and emotional problems (CBCL). The information obtained from children as well as from parental perspective will allow more extensive models on mechanisms of change.

Beyond psychometric instruments some well-established psychophysiological methods will be used. Assessment of the heart rate variability under mental stress conditions (Parametric Go/No-Go test) and measuring of cortisol awakening response (CAR) are used to study the function of autonomic nerve system and stress-level/tolerance of the study population.

The investigators hypothesize:

1. a significant decrease in number of days with pain/discomfort in both intervention groups (GDH, NS) as compared to the control group (active waiting-list control group)
2. that both types of intervention lead to an increase of quality of life and decrease of pain duration, intensity and pain-related disability as compared to the control group.
3. a decrease of physiological stress parameters (as measured by heart rate variability [HRV] analysis, cortisol awakening response [CAR]) in both intervention groups as compared to the control group, but more prominent in GDH group.

The data of this pilot study will be used for further projects where the most promising intervention and research parameters will be investigated more detailed in a larger sample.

Current study is regarded as a pilot and is conducted in order to obtain information about the efficacy of GDH and probiotic intervention in children with IBS or FAP as compared to reference group. Based on our previous studies and data of literature the investigators expect to see moderate effect power of the primary outcome measure (η²~.06). In order to detect a 50% improvement of symptoms during 4 week treatment with 80% power, assuming α=.05 and using a 2 x 3 repeated measure design for the main analysis, 51 participants should be included in the study. Taking into account possible dropouts the investigators plan to recruit 60 children (20 children per group).

Short description of study protocol: Parents that are interested in the study after a first contact with the investigators will receive detailed informations about the study and a short anamnestic questionnaire. After returning it they will be invited together with their children for the diagnostic appointment ("Visit I"). Inclusion into the study will be made based on the results of anamnestic interview as well as based on the reports from the responsible gastroenterologist regarding exclusion of other possible reason for the symptoms (including organic disorder, e.g. Celiac disease). Participants and their parents will also receive all necessary information about goals of the study and methods used in the study as well as about possible health risks from applied interventions. Informed consent is to be signed prior inclusion in the study. After inclusion, children and parents will be asked not to change any currently used medications or to undertake another treatment, as well as not to change usual habits until the end of the follow-up period.

Participants will be filling in diaries that will question about their symptoms once a day.

During the first two weeks ("run-in period") participants will only be keeping their symptom diaries. This data will be used in later analysis as "baseline" data for comparison with any changes that will occur due to intervention. The week three and four are regarded as "wash-out period": participants will be instructed to stop answering questions in diaries. The investigators hypothesize that this will reduce the effect of self-monitoring when the treatment starts.

At the end of week four, children will be randomized into one of three groups: based on computer generated table of random numbers each participant will be allocated either to a group practicing a gut-directed hypnosis or receiving a probiotic for the next four weeks (SymbioLact B) or reference group (only symptom diaries). Participants are randomized with an aspect ratio 1:1:1. Children will continue to keep the symptom diaries for another two weeks (week 9 and 10) and will return them to the investigators during "Visit II" at the end of 10th week.

Visits I and II will also be used to collect psychometric data from children and their parents as well as psychophysiological measures (HRV). Saliva samples should be collected at home: participants will be provided with appropriate collection tubes as well as with detailed instructions on how to collect, store and deliver samples to the investigation site. Baseline saliva samples should be collected inside the first week and during week 10 (in a morning before Visit II).

For ethical reasons, a second intervention can be chosen freely by the family after the follow-up period.

Risks of the study: A systematic review and meta-analysis of randomized clinical trials about the effects of probiotic in children with pain-related FGID as well as RCTs report seldom or no adverse effects from probiotics. If appeared - most often in a form of gastroenteritis and vomiting - the adverse effects were comparable to those in a placebo group. Based on previous studies of our group we expect no adverse events from gut directed hypnosis. All adverse events in any group will be documented and reported.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 17
* participants should fulfill following criteria for functional abdominal pain (FAP) or irritable bowel syndrome (IBS) according to Rome III Consensus
* medical report from a gastroenterologist about absence of an organic reason for the gastrointestinal complaints

Exclusion Criteria:

* organic reason for abdominal pain is diagnosed (e.g. celiac disease, inflammable bowel diseases)
* children fulfill criteria for abdominal migraine
* other acute or chronic disorders of the gastrointestinal, cardiovascular or peripheral nervous system are present
* inability to follow instructions

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in number of days with pain/discomfort | baseline, at week 10 and at 3 months follow-up

SECONDARY OUTCOMES:
Change in parental report on gastrointestinal symptoms (Abdominal Pain Index (API)) | baseline, at week 10 and at 3 months follow-up
Change in pain related disability (Pediatric Pain Disability Index (P-PDI)) | baseline, at week 10 and at 3 months follow-up
Change in somatic complaints (Children's Somatization Inventory (CSI)) | baseline, at week 10 and at 3 months follow-up
Change in health-related quality of life (KINDL-R Questionnaire) | baseline, at week 10 and at 3 months follow-up
  The KINDL-R is a generic instrument for assessing Health-Related Quality of Life in children and adolescents
Change in pain-related coping (Pediatric Pain Coping Inventory (PPCI)) | baseline, at week 10 and at 3 months follow-up
Change in emotional and behavioural problems (Child Behaviour Checklist (CBCL)) | baseline, at week 10 and at 3 months follow-up
Change in heart rate variability | baseline and at week 10
Change in cortisol awakening response (amount of cortisol in saliva, nmol/l) | baseline and at week 10
Change in self-reported pain intensity (Visual Analog Scale) | baseline, at week 10 and at 3 months follow-up
Change in self-reported pain duration (hours per day) | baseline, at week 10 and at 3 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marco D Gulewitsch, PhD, Principal Investigator — Eberhard Karls University, Tübingen, Germany
Locations (1):
- University Clinic, Tübingen, Germany

REFERENCES:
- [Background] Chitkara DK, Rawat DJ, Talley NJ. The epidemiology of childhood recurrent abdominal pain in Western countries: a systematic review. Am J Gastroenterol. 2005 Aug;100(8):1868-75. doi: 10.1111/j.1572-0241.2005.41893.x. PMID 16086724
- [Background] Schlarb AA, Gulewitsch MD, Bock Genannt Kasten I, Enck P, Hautzinger M. Recurrent abdominal pain in children and adolescents - a survey among paediatricians. Psychosoc Med. 2011 Mar 28;8:Doc02. doi: 10.3205/psm000071. PMID 21468324
- [Background] Chitkara DK, van Tilburg MA, Blois-Martin N, Whitehead WE. Early life risk factors that contribute to irritable bowel syndrome in adults: a systematic review. Am J Gastroenterol. 2008 Mar;103(3):765-74; quiz 775. doi: 10.1111/j.1572-0241.2007.01722.x. Epub 2008 Jan 2. PMID 18177446
- [Background] Campo JV, Di Lorenzo C, Chiappetta L, Bridge J, Colborn DK, Gartner JC Jr, Gaffney P, Kocoshis S, Brent D. Adult outcomes of pediatric recurrent abdominal pain: do they just grow out of it? Pediatrics. 2001 Jul;108(1):E1. doi: 10.1542/peds.108.1.e1. PMID 11433080
- [Background] Tack J, Fried M, Houghton LA, Spicak J, Fisher G. Systematic review: the efficacy of treatments for irritable bowel syndrome--a European perspective. Aliment Pharmacol Ther. 2006 Jul 15;24(2):183-205. doi: 10.1111/j.1365-2036.2006.02938.x. PMID 16842448
- [Background] Sandhu BK, Paul SP. Irritable bowel syndrome in children: pathogenesis, diagnosis and evidence-based treatment. World J Gastroenterol. 2014 May 28;20(20):6013-23. doi: 10.3748/wjg.v20.i20.6013. PMID 24876724
- [Background] Korterink JJ, Ockeloen L, Benninga MA, Tabbers MM, Hilbink M, Deckers-Kocken JM. Probiotics for childhood functional gastrointestinal disorders: a systematic review and meta-analysis. Acta Paediatr. 2014 Apr;103(4):365-72. doi: 10.1111/apa.12513. Epub 2014 Jan 7. PMID 24236577
- [Background] Tabbers MM, Chmielewska A, Roseboom MG, Crastes N, Perrin C, Reitsma JB, Norbruis O, Szajewska H, Benninga MA. Fermented milk containing Bifidobacterium lactis DN-173 010 in childhood constipation: a randomized, double-blind, controlled trial. Pediatrics. 2011 Jun;127(6):e1392-9. doi: 10.1542/peds.2010-2590. Epub 2011 May 23. PMID 21606153
- [Background] Banaszkiewicz A, Szajewska H. Ineffectiveness of Lactobacillus GG as an adjunct to lactulose for the treatment of constipation in children: a double-blind, placebo-controlled randomized trial. J Pediatr. 2005 Mar;146(3):364-9. doi: 10.1016/j.jpeds.2004.10.022. PMID 15756221
- [Background] Gulewitsch MD, Muller J, Hautzinger M, Schlarb AA. Brief hypnotherapeutic-behavioral intervention for functional abdominal pain and irritable bowel syndrome in childhood: a randomized controlled trial. Eur J Pediatr. 2013 Aug;172(8):1043-51. doi: 10.1007/s00431-013-1990-y. Epub 2013 Apr 9. PMID 23568514